CLINICAL TRIAL: NCT06953921
Title: Correlation Between Serum Albumin Level and Severity of Hepatic Encephalopathy in Patients With Chronic Liver Disease in Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Kerelos Latif sweha, Internal medicine resident, Sohag University
Other Study IDs: Soh-Med--25-3-02MS
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum albumin ALT AST
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assess the correlation between serum albumin levels and the severity of hepatic encephalopathy in patients with chronic liver disease.

assess the impact of albumin level on clinical course and outcomes of HE.

DETAILED DESCRIPTION:
sample size calculation will be performed based on anticipated incidence rates of HE and variability in serum albumin levels, aiming for a study population of 100-150 patients to achieve adequate statistical power.

- All patients included in the study will be subjected to : Glasgow Coma Scale (GCS) score. Clinical Assessment: Baseline evaluation of patients to confirm chronic liver disease diagnosis and determine clinical characteristics.

History of prior episodes of HE, presence of ascites, variceal bleeding, and other complications of chronic liver disease .

Age, gender, etiology of cirrhosis (e.g., viral hepatitis, alcohol), comorbid conditions (e.g., diabetes, hypertension)

* Laboratory investigation :

Serum albumin level AST ALT Total bilirubin and direct CBC Serum creatinine Proth time and concetntration

ELIGIBILITY:
Inclusion Criteria:

* patients aged >18 years.
* Confirmed chronic liver disease (by imaging ,
* liver function tests , and clinical history).
* Diagnosed with hepatic encephalopathy based on clinical criteria.
* Patients able to provide informed consent.

Exclusion Criteria:

* Patients age less than 18 years old
* Acute liver failure.
* Chronic renal failure on dialysis.
* Pregnant women.
* Patients with active malignancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: sample size calculation will be performed based on anticipated incidence rates of HE and variability in serum albumin levels, aiming for a study population of 100patients to achieve adequate statistical power.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
assess the correlation between serum albumin levels and the severity of hepatic encephalopathy in patients with chronic liver disease. | 6 months
  assess the impact of albumin level on clinical course and outcomes of HE.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided